CLINICAL TRIAL: NCT06298838
Title: Perioperative Assessment of Intraoperative Margins and Lymph Node Invasion Using High-resolution 18F-PSMA-PET-CT in Prostate Cancer: a Pilot Study
Brief Title: High-resolution Intra-operative PSMA PET-CT in Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giorgio Gandaglia, Assistant Professor, IRCCS San Raffaele
Other Study IDs: XEOS study
Record Dates: First submitted 2024-02-20; First posted 2024-03-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: AURA10® Specimen PET/CT imager — The AURA10 PET-CT specimen imager detects and measures the electron density distribution of a specimen and the radiotracer distribution within a specimen. The function of the system is to acquire and visualize PET and CT images of a specimen, based on which a healthcare professional can rapidly verify whether the correct tissue has been resected. It can be used in any condition that requires resection surgery to visualize the resected specimen. The device is automated and semi-quantitative, i.e., qualitative regarding visualization of structure and radiotracer distribution and quantitative regarding tissue density (Hounsfield units) and radiotracer uptake in the specimen (Bq/ml). The type of specimen required is resected tissue from a patient undergoing resection surgery.

SUMMARY:
This is a Single-center, diagnostic open-label prospective, pilot study in a total of 10 patients affected by Prostate cancer (PCa) with a risk of lymph node invasion (LNI) higher than 5% and candidates for a robot-assisted radical prostatectomy (RARP) with an extended pelvic lymph node dissection (ePLND) .

The aim of the trial is to evaluate the feasibility and accuracy and clinical value of a novel high-resolution perioperative PET-CT-scan for intraoperative margin and lymph node invasion assessment, after 18F-PSMA injection, using histopathology as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Male patient, 18 years of age or older.
2. Patient is confirmed with high risk prostate cancer.
3. Patient is indicated to undergo radical prostatectomy and ePLND.
4. Patient is estimated compliant for study participation by the investigator.
5. Patient has freely given his/her informed consent to participate in this study.

Exclusion Criteria:

1. Patient has general or local contra-indications for radical prostatectomy.
2. Patient has active viral or fungal infection.
3. Patient previously received radiotherapy of the prostate.
4. Patient participated in other clinical studies with radiation exposure of more than 1 mSv in the past year.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Prostate cancer (PCa) with a risk of lymph node invasion (LNI) higher than 5% and candidates for a robot-assisted radical prostatectomy (RARP) with an extended pelvic lymph node dissection (ePLND) according to the European Association of Urology (EAU) guidelines.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To investigate the performance characteristics (sensitivity and specificity) of a novel high-resolution perioperative PET-CT-scan for intraoperative margins and lymph node invasion assessment after 18F-PSMA using histopathology as the gold standard | 1 YEAR

SECONDARY OUTCOMES:
Reporting positive lymph nodes detection rate at intraoperative imaging after 18-PSMA injection | 1 YEAR

IPD SHARING:
Plan to Share IPD: Undecided